CLINICAL TRIAL: NCT04593901
Title: Protecting Home Healthcare Workers: An Interactive Video-based App to Coach Workers Through Challenging Health and Safety-related Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Amy Darragh, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GRT00054864
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Occupational Exposure
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Study is pre-intervention that uses a participatory, iterative approach to develop an app for use in subsequent intervention studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video and App Review (Other): Single arm study in which home healthcare workers review and provide feedback on scripts and/or videos and on the usefulness, usability, and desirability of an interactive app in an iterative, participatory manner.
  Interventions: Behavioral: Video and App Review

INTERVENTIONS:
Behavioral: Video and App Review — Scenario Review: The scripts and/or videos will be iteratively reviewed by individual and small groups of home healthcare personnel using Zoom, Microsoft Teams, or similar. The participants will review scripts and/or recordings of the scripts and discuss how well each situation has been represented, how to improve it, and whether it is applicable in their agency.
  App Review: Following review of the scenarios, participants will review the smartphone app currently under development, including the control buttons, their placements, and other features of the screen interface. The first 9-12 participants (approximately) will be asked to provide feedback on the app's layout, control locations, and overall appearance. Once suggested changes have been made, the app will then be reviewed by the remaining participants for final review and usability assessment.

SUMMARY:
This project will create a video-based app that empowers home healthcare workers to communicate with clients and their families about managing health and safety hazards in client homes. Using a participatory approach, home healthcare workers will 1) review and revise video scripts and recordings that demonstrate effective and less effective communication strategies when talking to clients, families, and other stakeholders about health and safety hazards and 2) contribute to the creation and review of an interactive app that they perceive to be useful, usable, and desirable.

DETAILED DESCRIPTION:
This project includes two of three original aims. The first aim (Aim 1), already completed, created scripts based on real-world scenarios regarding speaking with clients and families about health and safety hazards in their homes.

Based on the data from Aim 1, the research team has prepared scripts describing each scenario. Each scenario includes two to three different approaches that represent successful, less successful, and/or unsuccessful examples of communicating about solving difficult or complex health and safety challenges. Each scenario includes a short introductory statement about the context of the scenario and two to three subsequent scripts and/or recordings that demonstrate the different communication approaches. Scenarios with successful communication strategies present the approach and outcomes that are consistent with best practices for HHW's in a given situation.

In Aims 2 and 3, participants will participate in either an individual or group interview using Zoom, Teams, or similar. They will review scripted scenarios and, as they are developed, video recordings based on the scripted scenarios. They will answer questions about the relevance of the information, how realistic the dialogue is, the usefulness of the information, and changes/improvements they would make. In addition, participants will review an app designed to allow users to select the videos they wish to view, and view successful, less successful, and unsuccessful communication approaches and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Home healthcare worker (including clinical, professional, and administrative staff)
* 18+ years of age
* 6 months of home healthcare experience
* access to computer/tablet/smartphone

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Usefulness, Usability, Desirability Assessment | The UUD Assessment is administered once 1 day a participant has reviewed the app in order to assess overall usability. It is completed only once by each participant.
  This flexible and individualized instrument uses a 5 point-Likert scale to assess whether the app was useful, easy to use, and appealing

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan as of yet given small n and qualitative nature of data.